CLINICAL TRIAL: NCT01244971
Title: Effect of Exercise Training - Alone or in Combination With Acarbose - on Clinical and Metabolic Factors, and Studies of Cellular and Moleculargenetic Factors, in Type 2 Diabetes.
Brief Title: Exercise and Acarbose in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government); Bayer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNR 03-539
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2010-11-22 (Estimated); Status verified 2003-12

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acarbose; Exercise

ARMS (3):
- Acarbose (Active Comparator)
  Interventions: Drug: Acarbose
- Exercise (Active Comparator)
  Interventions: Behavioral: Exercise
- Exercise + Acarbose (Experimental)
  Interventions: Other: Exercise + Acarbose

INTERVENTIONS:
Drug: Acarbose — 100mg, 3 times daily
  Arms: Acarbose
Behavioral: Exercise — Moderate combined exercise, 50 minutes 3 times per week
  Arms: Exercise
Other: Exercise + Acarbose — See respective monotherapy description
  Arms: Exercise + Acarbose

SUMMARY:
The purpose of this study is to investigate the impact of exercise training, Acarbose, and the combination of exercise and Acarbose on glycemic control, body composition, insulin sensitivity and other cardiovascular risk markers in type 2 diabetes. Further, muscle biopsies will be obtain to study gene expression. Our hypothesis is that the combination therapy will be superior to monotherapy with exercise or Acarbose.

ELIGIBILITY:
Inclusion Criteria: Men and women, diagnosis of type 2 diabetes established since at least three months, treatment with diet or maximum one oral anti-diabetic drug, GHb < 8.5 %, age 45 - 60 years, BMI 25 - 30 kg/m2, no participation in any regular exercise program.

-

Exclusion Criteria: Unable to perform exercise, significant GI-disease, severe heart-disease, renal failure

-

Ages: 45 Years to 60 Years | Sex: All
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2004-01; Primary Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Glycemic control | 12 weeks
  Glycated A1c

CONTACTS AND LOCATIONS:
Overall Officials: Suad Efendic, Professor, Study Chair — Dpt of Molecular Medicine and Surgery, Karolinska Institutet, Stockholm, Sweden
Locations (1):
- Enheten för Metabol Kontroll, Endokrinkliniken, Karolinska University Hospital, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Result] Wagner H, Degerblad M, Thorell A, Nygren J, Stahle A, Kuhl J, Brismar TB, Ohrvik J, Efendic S, Bavenholm PN. Combined treatment with exercise training and acarbose improves metabolic control and cardiovascular risk factor profile in subjects with mild type 2 diabetes. Diabetes Care. 2006 Jul;29(7):1471-7. doi: 10.2337/dc05-2513. PMID 16801564